CLINICAL TRIAL: NCT04274049
Title: A Phase III, Double-Blind, Randomized, Placebo-Controlled, Multicenter Study to Assess the Safety and Efficacy of NL003 in Subject With Critical Limb Ischemia（Rutherford 5）
Brief Title: Safety and Efficacy Study Using Gene Therapy for Critical Limb Ischemia (NL003-CLI-III-2)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Beijing Northland Biotech. Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NL003-CLI-III-2; CTR20190750 (Other: National Medical Products Administration（China）chinadrugtrials.org.cn)
Record Dates: First submitted 2020-01-18; First posted 2020-02-18 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Arterial Occlusive Disease; Ischemia; Ulcers; Peripheral Vascular Disease
Keywords: HGF; Gene; Critical Limb Ischemia
MeSH Terms: conditions — Arterial Occlusive Diseases; Ischemia; Ulcer; Peripheral Vascular Diseases; Chronic Limb-Threatening Ischemia | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- investigational produc (Experimental): Patients in this treatment group will receive 8mg NL003 respective in D0、14、28
  Interventions: Genetic: NL003
- Placebo (Placebo Comparator): Patients in this group will receive normal saline respective in D0、14、18
  Interventions: Other: Normal Saline

INTERVENTIONS:
Genetic: NL003 — Day 0: 8mg of NL003 (32 injections of 0.5ml of NL003) Day 14: 8mg of NL003 (32 injections of 0.5ml of NL003) Day 28: 8mg of NL003 (32 injections of 0.5ml of NL003)
  Other Names: HGF plasmid; pCK-HGF-X7
  Arms: investigational produc
Other: Normal Saline — Day 0: 16ml of Normal Saline (32 injections ) Day 14: 16ml of Normal Saline (32 injections ) Day 28: 16ml of Normal Saline (32 injections )
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate whether intramuscular injections of NL003 into the calf is safe and effective in the treatment of critical limb ischemia

DETAILED DESCRIPTION:
Management of CLI process consumes a significant amount of healthcare resources,and the new therapeutic approaches are required.

Hepatocyte growth factor (HGF) has been shown to be a potent angiogenic growth factor stimulating the growth of endothelial cells and migration of vascular smooth muscle cells. Because of its pluripotent capabilities, increasing the availability of HGF in ischemic tissues to achieve therapeutic angiogenesis has been a growing area of research.

This study will use NL003, which is a DNA plasmid that contains novel genomic cDNA hybrid human HGF coding sequence (HGF-X7) expressing two isoforms of HGF, HGF 728 and HGF 723. As there are currently no approved drugs that can reverse CLI and as most patients have exhausted surgical and endovascular intervention options, inducing angiogenesis in the affected limb with NL003 may result in an increase in tissue perfusion, which, in turn improve wound healing, reduce pain and improve limb salvage rates.

ELIGIBILITY:
Inclusion Criteria:

* 1. At the age of 20 and 80 (at the time of signing the informed consent), both male and female.

  2. According to DSA or CTA, patients diagnosed with lower limb arterial ischemic disease based on the medical history and clinical manifestations and with Rutherford grade 5 (with ulcer) must meet the substandardProspective.(if both limbs of the subject suffer from lower limb arterial ischemic disease, it is up to the investigator to select one limb for the study.)Resting ankle systolic pressure (dorsal foot artery or posterior tibial artery) ≤70mmHg or ABI≤0.5 or TcPO2 < 30mmHg;In the first 3 months after randomized inclusion, DSA or CTA confirmed severe stenosis (≥70%) or occlusion of superficial femoral artery or popliteal artery or inferior knee artery.

  3. Patients with chronic lower limb arterial ischemia complicated with ulceration also met the following requirements: when signing the informed consent, the ischemic ulcer of the artery lasted at least 2 weeks;When signing the informed consent, the area of a single ulcer is no more than 10cm2;If there are multiple ulcers in the affected limb selected at the time of signing the informed consent, the total number of ulcers shall not exceed 3.Basic ulcer care (according to standard ulcer care procedure) should be maintained during the test to avoid aggravation of infection.The ulcer did not expose bone or joint capsule.If there is gangrene, only partial toe gangrene.

  4. Agreed to use the basic treatment drugs as required during the test, and kept a complete record of the subjects' diaries on time. The compliance of the basic treatment drugs and the subjects' diaries during the screening period was ≥70%.

  5. Agree to use appropriate contraceptive measures during the experiment;Female subjects of reproductive age, blood pregnancy test negative.

  6. Signed informed consent.

Exclusion Criteria:

* 1. Patients with acute lower limb ischemia or acute exacerbation of chronic lower limb ischemia.

  2. Vascular reconstruction (bypass or intravascular therapy) or sympathetic resection or amputation was performed within 4 weeks prior to the signing of the informed consent.

  3. Due to the surgical operation, the patient was still in the postoperative risk period, and the researcher judged that it was not suitable for the participant.

  4. Main-iliac artery stenosis ≥70%.

  5. Severe limb infection (cellulitis, osteomyelitis, etc.), distal fascia or bone exposure were observed.

  6. Cardiac function NYHA class belongs to Ⅳ grading standards (see appendix 1).

  7. Cerebral infarction, cerebral hemorrhage, myocardial infarction or unstable angina pectoris occurred within 3 months before signing the informed consent.

  8. Refractory hypertension (systolic blood pressure ≥180mmHg or diastolic blood pressure ≥110mmHg when taking three or more antihypertensive drugs).

  9. Proliferative retinopathy and retinopathy examination is not available.

  10. Inability to accurately describe symptoms and emotions.

  11. Severe liver disease with uncompensated cirrhosis, jaundice, ascites or hemorrhagic varices.

  12. Current recipients of immunosuppressants or chemoradiotherapy.

  13. Anti-hiv antibody positive, anti-hepatitis c antibody positive and hepatitis b surface antigen positive (if the subject is HBsAg positive and HBV DNA in peripheral blood is combined, the researcher believes that the subject's chronic hepatitis b is stable and will not increase the risk of the subject, the subject can be selected).

  14. Results of laboratory examination during screening period: hemoglobin < 80g/L, white blood cell count < 3.0×109/L, platelet < 75×109/L, upper limit of normal AST or ALT >, upper limit of normal serum creatinine > was 3 times, or other laboratory examination indicators showed abnormalities that researchers thought might affect the evaluation of test results.

  15. Poor blood glucose control after treatment (glycosylated hemoglobin > 10%).

  16. Previously diagnosed with malignant tumor, or any of the following test results determined by the investigator to be at risk of tumor: fecal occult blood test;Chest X-ray examination or chest CT examination;Alpha-fetoprotein (AFP), carcinoembryonic antigen (CEA) and ca19-9;Male subjects, prostate specific antigen test (PSA, free PSA);Female subjects: cervical smear (Pap), mammography/b-ultrasound, ca-125;The investigators determined that additional tests were necessary to eliminate the tumor risk.

  17. In the opinion of the investigators, patients with comorbidities that affect safety and efficacy evaluation, or those with a predicted survival of less than 12 months.

  18. Frequent drinkers within the 12 months prior to the signing of the informed consent, i.e., those who drank more than 14 units of alcohol per week (1 unit =360 mL beer or 45 mL alcohol of 40% spirits or 150 mL wine) or substance abusers.

  19. Participate in other clinical trials within 3 months before signing the informed consent.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2019-08-28 (Actual); Primary Completion 2023-12-23 (Actual); Study Completion 2023-12-23 (Actual)

PRIMARY OUTCOMES:
Percentage of ulcer complete healing | Day180
  1.At D180 visit, subjects intended to observe the healing of all arterial ischemic ulcers in the limb;2.Ulcer healing criteria: skin epidermal cell regeneration without secretion.

SECONDARY OUTCOMES:
The time when the ulcer finally heals completely | Day14,Day28,Day60,Day90,Day120,Day180
  The time between the first use of the study drug and the final full healing of the ulcer.
Percentage of cases with ulcer area reduced by ≥50% from baseline | Day180
  The ulcer area at the last visit was 50% less than the baseline case percentage.
Percentage of new ulcer or gangrene cases | Day14,Day28,Day60,Day90,Day120,Day180
  The percentage of new ulcer or gangrene cases after use of the study drug.
Rate of complete disappearance of pain | Day180
  Rate of complete disappearance of pain.
Percentage of cases with a 50% reduction in pain score from baseline | Day180
  A 50% reduction in pain score from baseline at the last visit.
Changes in pain score from baseline | Day14,Day28,Day60,Day90,Day120,Day180
  The severity of critical Limb ischemia was assessed by Rutherford grading at screening, D14, D28, D60, D90, and D180, respectively.
Changes in quality of life scores from baseline | Day14,Day28,Day60,Day90,Day120,Day180
  The quality of life score questionnaire was conducted to evaluate the subjective perception of Critical Limb Ischemia, including the subjects' perception of quality of life, health, or other aspects of life.
Changes in Rutherford grading from baseline | Day14,Day28,Day60,Day90,Day120,Day180
  The severity of critical Limb ischemia was assessed by Rutherford grading at screening, D14, D28, D60, D90, and D180, respectively.
Changes to the ABI from the baseline | Day60,Day90,Day120,Day180
  Ankle-brachial index (ABI) refers to the ratio of systolic blood pressure of the anterior tibial artery (dorsal foot artery) or posterior tibial artery to the systolic blood pressure of the brachial artery.Participants were tested for ankle-brachial index (ABI).
The percentage of patients who undergo revascularization (open surgery or interventional therapy) has a high amputation rate of mortality | Day180
  The percentage of patients who undergo revascularization (open surgery or interventional therapy) has a high amputation rate of mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Changwei Liu, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (21):
- China (21):
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Zhongshan Hospital Xiamen University, Xiamen, Fujian
  - Zhangzhou Municipal Hospital of Fujian Province, Zhangzhou, Fujian
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - Xuzhou Mining Group General Hospital, Xuzhou, Jiangsu
  - The First Affiliated Hospital of Zhengzhou University, Changchun, Jilin
  - Affiliated Hospital of Inner Mongolia Medical University, Baotou, Neimenggu
  - Chifeng Municipal Hospital, Chifeng, Neimenggu
  - Affiliated Hospital of Shandong University of Traditional Chinese Medicine, Jinan, Shandong
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Qingdao Hiser Hospital Affiliated of Qingdao University（Qingdao Traditional Chinese Medicine Hospital）, Qingdao, Shandong
  - Fudan University Affiliated Pudong Medical Center, Shanghai, Shanghai Municipality
  - Shanghai 9th People's Hospital Affiliated to Shanghai JiaoTong University, School of Medicine;, Shanghai, Shanghai Municipality
  - Shanxi Provincial People's Hospital, Taiyuan, Shanxi
  - First Affiliated Hospital of Xi 'an Jiaotong University, XiAn, Shanxi
  - The First Affiliated Hospital，Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
  - zhongshan Hospital Affiliated of Dalian University, Dalian